CLINICAL TRIAL: NCT06749574
Title: Effectiveness of Stability Ball Training, Dead Bug Exercises, and Their Combination on Reducing Specific Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/774
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Radiculopathy Lumbar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stability ball Training (Active Comparator)
  Interventions: Diagnostic Test: stability ball exercises
- Dead bug training: (Experimental)
  Interventions: Diagnostic Test: dead bug exercise
- Combined Group (Active Comparator)
  Interventions: Combination Product: Combined Groupo

INTERVENTIONS:
Diagnostic Test: stability ball exercises — articipants in the first group performed stability ball exercises designed to enhance balance, core stability, they were introduced to the stability ball with instructions on maintaining proper posture, alignment, and safety to prevent injuries. The program included exercises such as the Stability ball bridging, stability ball bird dog and stability ball pelvic tilts were included to activate the lower abdominal muscles and glutes through gentle, controlled movements
  Arms: Stability ball Training
Diagnostic Test: dead bug exercise — The second group focused on dead bug exercises, Participants performed exercises such as extending one arm and the opposite leg while lying on their backs, ensuring their spine remained neutral and their lower back stayed pressed into the floor. Variations included alternating opposite arm and leg movements and holding the extended position to increase the challenge and enhance core stability. These exercises were performed slowly to maintain control and improve movement precision over the eight-week period
  Arms: Dead bug training:
Combination Product: Combined Groupo — The third group combined stability ball and dead bug exercises for a comprehensive training approach targeting both core stability and balance. Participants alternated between dead bug exercises, which required controlled arm and leg extensions while lying on their backs, and stability ball exercises such as the ball with bridging and bird dog. Throughout the eight weeks, participants were encouraged to maintain proper posture, alignment, and a neutral spine during all activities to ensure safety and effectiveness
  Arms: Combined Group

SUMMARY:
This study is a single-blinded, randomized controlled trial (RCT) focused on individuals aged 30 to 50 with acute specific low back pain (lumbar radiculopathy). Participants will be divided into three groups: one performing stability ball exercises, one doing dead bug exercises, and the third group combining both types of exercises.

DETAILED DESCRIPTION:
The study aims to assess the effectiveness of these regimens in reducing pain and improving quality of life. The trial will be conducted at Sheikh Zayed Hospital and Alara Health Care Clinic, with simple random sampling used to assign participants. The study will run for 6 months, with follow-up assessments at 1, 4, and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 30 to 50 years with a specific diagnosis of acute lumbar radiculopathy lasting less than three months but severe enough to impair daily activities were included in the study.
* They were required to provide informed consent and agree to adhere to the study procedures,
* including attending sessions and completing evaluations. Eligibility was limited to those without other physical conditions, such as joint replacements or fractures,
* that could interfere with the ability to perform stability ball or dead bug exercises. Individuals who had participated in similar therapeutic exercises, such as stability ball training or core strengthening, within the last six months were excluded to ensure the results reflected the intervention's impact rather than prior training effects.

Exclusion criteria:

* included participants with severe musculoskeletal or cardiovascular disorders, such as spinal surgery, herniated discs, scoliosis, fractures, or osteoarthritis, due to the potential risks associated with exercise.
* Pregnant women were excluded as balance-related activities, like stability ball exercises, could pose safety concerns. Individuals using pain medications, particularly opioids or muscle relaxants, were excluded to avoid interference with exercise performance or altered pain perception.
* Participants who had undergone back surgery within the last six months, or those currently undergoing other physical therapy or treatments for back pain, such as physiotherapy or chiropractic care, in the previous month were also excluded

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 12 Months
  The VAS (Visual Analog Scale) is used for pain assessment. It consists of a vertical line, with the words 'No pain' at the bottom end corresponding to a VAS of 0, and 'Worst pain possible' at the top end corresponding to a VAS of 10.
SF-12 (Short Form 12-Item Health Survey) | 12 Months
  widely used questionnaire designed to assess health-related quality of life. It is a concise version of the SF-36, retaining 12 carefully selected questions that measure physical and mental health domains. The SF-12 evaluates eight health components: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional health problems, and mental health.Responses from the SF-12 are used to generate two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). These scores provide a quantitative measure of an individual's physical and mental well-being, respectively. The PCS focuses on physical health aspects like mobility and pain, while the MCS emphasizes emotional health and social functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Zayed Hosp and Alara Health Care Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No